# 1 Hypolipidemic and Antioxidant Capacity of Spirulina and Exercise

2 NCT number: NCT02837666.

3 Date: April 27, 2017

4 Responsible: Dr. Arnulfo Ramos Jiménez

5 Autonomous University of Ciudad Juárez, México

6 e-mail: aramos@uacj.mx

#### 7 Abstract

- 8 **Introduction:** In order to reduce cardiovascular diseases risk factors, a healthy
- 9 diet must include dietary antioxidants from different sources (e.g. Spirulina
- 10 maxima) and regular practice of exercise should be promoted.
- 11 There is a little evidence from animal studies that *Spirulina maxima* and exercise,
- decreases cardiovascular diseases risks factors. However, very few studies have
- proven the independent or synergistic effect of *Spirulina maxima* plus exercise in
- humans. Therefore, this study pretends to address this independent and
- synergistic effect in overweight and obese subjects participating in a systematic
- physical exercise program at moderate intensity on general fitness, plasma lipid
- profile and antioxidant capacity in overweight and obese subjects.
- 18 **Methods and analysis:** Through a randomized, double-blind, placebo-controlled,
- and a counterbalanced crossover study design, eighty healthy overweight, and
- 20 obese subjects will be evaluated during a twelve-week isoenergetic diet,
- 21 accompanied by 4.5 g a day of *Spirulina maxima* intake and/or a physical
- 22 systematic exercise program at moderate intensity. Body composition, oxygen
- uptake, heart rate, capillary blood lactate, plasma concentrations of triacylglycerols,
- total, low and high-density lipoprotein cholesterol, antioxidant status, lipid oxidation,
- 25 protein carbonyls, superoxide dismutase, catalase, glutathione, glutathione
- peroxidase, glutathione reductase, and paraoxonase will be assessed.
- 27 **Ethics and dissemination:** This study and all the procedures have been approved
- by the Universidad Autonoma de Ciudad Juarez Bioethics Committee. Moreover,

- 29 findings will be disseminated through peer-reviewed journals, national and
- 30 international conferences.
- Trial registration number: ClinicalTrials.gov: NCT02837666.
- 32 **Keywords:** Spirulina, dyslipidemias, oxidative stress, exercise, body fat,
- 33 antioxidant.

# 34 Strengths and limitations of this study

- Working with obese people, one of the main risk factors for cardiovascular
   diseases.
- This study can be extrapolated to different populations.
- Double-blind randomized controlled trial.
- There are not possible limitations to perform all the procedures described in the present paper.

# Background

- 42 Cardiovascular diseases (CVD) are the leading causes of death worldwide. Each
- year, 17.5 million people die because of these diseases <sup>1</sup>. Dyslipidemias are a
- 44 predisposing factor for CVD and are characterized by high concentrations of
- 45 triacylglycerols (TAG), total cholesterol (TC), low-density lipoproteins cholesterol
- (LDL-c), and low concentrations of high-density lipoproteins cholesterol (HDL-c)<sup>2</sup>.
- Besides dyslipidemias, oxidative stress (OxS) is also observed to rise in obesity <sup>3,</sup>
- 48 <sup>4</sup>, and it is also a predisposing factor for CVD <sup>5-8</sup>.

- 49 As a way to reduce OxS, dyslipidemias and the CVD incidence, it has been
- 50 proposed the intake of antioxidants that come from fruit and vegetable-rich diet or
- nutritional supplements, mainly by unprocessed foods <sup>9, 10</sup>. In this sense,
- 52 cyanobacterium *Spirulina* is an important source of antioxidants, currently
- associated with cardiovascular protection properties <sup>9, 11</sup>.
- For centuries, *Spirulina maxima* (*S. maxima*) has been cultivated and used as a
- 55 nutritional supplement due to its content of amino acids and essential fatty acids,
- vitamin C, vitamin E, tocopherols, and phycocyanins <sup>12</sup>. Recently, *S. maxima*
- 57 studies have focused in verifying the biological activity of its components, including
- 58 hypolipidemic and antioxidant effects <sup>13-15</sup>. However, most studies have been
- conducted in animal models, with only a few studies focused on the biological
- 60 effect in humans.
- Furthermore, it is known that the practice of systematic physical exercise
- ameliorates CVD risks <sup>10, 16</sup>; and it has been observed that also plays a role in OxS,
- especially physical exercise at high intensity (PEHI) <sup>17</sup>. PEHI considerably
- increases general metabolism, oxygen uptake (VO<sub>2</sub>), and mitochondrial activity;
- thus increasing the reactive oxygen species (ROS) production<sup>18</sup>. Instead, physical
- exercise of moderated intensity (PEMI) has the best protective effect exerted
- against CVD, mainly due to physiological adaptations, including the expression of
- antioxidant enzymes <sup>19</sup>, which stop the formation and propagation of ROS, and
- improving redox status of the organism <sup>20, 21</sup>.
- Algae and cyanobacteria have shown promising pharmacological properties
- providing health benefits and physical improvements <sup>22</sup>. These effects are

- attributed to their specific profile in bioactive compounds such as uncommon
- carotenoids, phenolic compounds, tocopherols besides their well-known content in
- vitamins and good quality proteins associated to their specific chemical structure
- and interaction with biological membranes <sup>23</sup>.
- In this sense, there is evidence that the cyanobacteria *Spirulina*, in addition to
- exercise, lower CVD risks. This was mainly observed in animal models <sup>24-26</sup>.
- However, no studies in humans under *Spirulina* and exercise experimental designs
- 79 proving these benefits have been reported yet. Therefore, the ISESE study will
- analyses the independent and synergistic effect of the intake of *S. maxima* with a
- PEMI on general fitness, plasma lipid profile, and redox status in overweight and
- 82 obese subjects.

# Methods/Design

# 84 Hypothesis

83

87

91

- 85 Spirulina maxima intake and a dosed physical activity program will improve lipids
- profile, general fitness and antioxidant status in overweight and obese subjects.

# Objectives

- The ISESE project's main objective is to demonstrate that ingestion of *S. maxima*
- and a dosed physical activity program will decrease, both independently and
- synergistically, some CVD risks in overweight and obese subjects.

# **Outcome measures**

- The primary outcome measure will be changes in the plasma lipid profile after a
- 93 six-week of treatment (plasma TAG, TC, HDL-c, and LDL-c by using standardized
- 94 enzymatic methods).
- The secondary outcome measure will be changes in general fitness (maximal
- oxygen uptake (VO<sub>2</sub> max), heart rate (HR), in onset blood lactate accumulation,
- and body fat mass); as well as changes in redox status (malondialdehyde (MDA),
- 98 protein carbonyls, paraoxonase (PON1), superoxide dismutase (SOD), catalase
- 99 glutathione (GSH), glutathione reductase (GR), and glutathione peroxidase (GPx).

# Participants' eligibility

100

109

- The inclusion criteria will be the age between 18 and 45 years old of both sexes:
- 40 overweight (Body mass index (BMI): 25-29.9 kg/m<sup>2</sup>) and 40 obese (BMI: >30
- kg/m<sup>2</sup>). The subjects' exclusion criteria will be: drinking more than 100 mL of
- alcohol a week, taking drugs and/or food or vitamin supplements, having a chronic
- disease, or having a physical or electrocardiographic injury that prevents them from
- engaging in any regular physical exercise. The elimination criteria will be that the
- program subjects' attendance will be lower than 80% and/or 20% change in their
- 108 body weight during study.

# Call to participation, ethics and safety procedures

- 110 University students of Ciudad Juarez, Mexico with overweight and obesity will be
- personally invited to participate. Participants will be informed of the purpose of the
- study, and of the physical, clinical and biochemical procedures, benefits, physical
- intensity tests, and risks, all before beginning the clinical trial. To guarantee the

good physical and mental health of the participants at the beginning of all the studies, a medical clinical laboratory study examination and an electrocardiography at rest tests will be performed. Noting that investigators are trained in cardiopulmonary reanimation and that the laboratory has the necessary communication tools and channels to perform emergency procedures. This study and all the procedures have been registered appropriately in ClinicalTrials.gov database (NCT02837666) and approved by the Bioethics Committee of the Universidad Autonoma de Ciudad Juarez (Supplementary files). That participants' acceptance formalized by means of written informed consent and their anonymity and confidentiality will be strictly enforced. This study will be conducted in compliance with the principles of the Declaration of Helsinki.

#### **Baseline measurements**

A day before beginning the treatment, subjects will visit the laboratory for baseline measurements. Body mass will be measured with subjects lightly dressed and barefoot in an electronic balance, and standing height with a stadiometer. Body fat percentage will be measured by plethysmography method (BodPod, USA), electric bioimpedance (in body 160, US), and by dual-energy X-ray absorptiometry (DXA) (Prodigy v6.8; GE Lunar, Milwaukee, WI) according to manual guidelines. Anthropometric parameters will be taken by the standardized method of the International Society for the Advancement of Kinanthropometry (ISAK), and according with ISAK Anthropometry Accreditation protocols <sup>27</sup>. Researchers are standardized in handling equipment and procedures. 

# Study design

The study consists of *S. maxima* treatment during 14 weeks in a randomized. double-blind, placebo-controlled, and counterbalanced crossover design, aimed to eliminate inter-individual bias as well as boosting the reliability of final results; moreover, this design is commonly used in clinical trials in order to have better results and conclusions <sup>28</sup>. Eligible participants (n= 80) will be divided into two groups, one with systematic practice of physical exercise (GEx) and other one without it (GNEx). The participants of each group will be randomized in equal proportions between S. maxima and placebo treatment, receiving either 4.5 g daily, in a non-transparent capsule during 12 weeks (6 weeks for the first treatment - 2 weeks of washout period - 6 weeks for the second treatment) (Figure 1). Before any reported allergic reaction occurs, the treatment will be discontinued. To maintain the overall quality and legitimacy of the clinical trial, code interruptions should occur only in exceptional circumstances when knowledge of the actual treatment is essential for further management of the participant. Investigators are encouraged to discuss with a Medical Advisor if they believe that unblinding is necessary. Unblinding should not necessarily be a reason for study discontinuation. A student outside the research team will feed data into the computer in separate datasheets, so that the researchers can analyze the data without having access to information about the allocation treatments, storing all the participants' files in numerical order in a safe and accessible place. The participants' files will be stored for a period of five years after the end of the study.

137

138

139

140

141

142

143

144

145

146

147

148

149

150

151

152

153

154

155

156

157

The sample size was determined by using the statistical program G\*Power  $^{29}$ , selecting a sample of 73 subjects with  $\alpha$  = 0.05 and p = 0.85. This sample will be fixed to 80 subjects in order to anticipate the possible desertions from the study.

# **Maximum intensity tests**

159

160

161

162

163

164

165

166

167

168

169

170

171

172

173

174

175

176

177

178

179

180

181

Each subject will participate in four stress tests performed at maximum intensity (MIT) during the study; during MIT record, consumed O<sub>2</sub> and produced CO<sub>2</sub> will be taken by a gas analyzer (Cortex MetaLyzer® 3B, Germany), HR with a Polar H7 sensor (Polar Electro, Lake Success, NY), and lactate in capillary blood samples will be assayed in a YSI 1500 Sport Lactate Analyzer (YSI Life sciences, OH, USA). The MIT protocol consists of using a cycle ergometer (Monark ergomedic 828 E; Monark exercise AB, 105 Vansbro, Sweden) initiating with a workload of 50-75 W with increments of 15-30 W every 3 min for until 15 min or when the subject could no longer pedal more than 40 revolutions/min, finishing the test when reaching 90-100 % of the maximum HR reserve; MIT will not be valid for less than 9 min (Figure 2). At the end of each increment load (3 min), capillary blood samples will be taken to determine lactate, and the physical perceived effort will be registered by using the Borg scale. Measurements of HR, glucose and blood pressure will serve to take care of the subject's health during each MIT. Before the first MIT, subjects will decide to be in the GEx or GNEx, and then they will be divided randomly for the treatment, which consists in a daily dosage of 4.5 g of Spirulina or placebo in capsules which will be recommended the subjects to consume them before each meal every day during six weeks. The day after the first supplementation period, subjects will come back to perform the second MIT

with identical conditions to the first one. The third MIT will be performed after a washout period of two weeks to remove the effects of treatment and avoid any possible delayed effect of *S. maxima* in the organism. The last MIT will be performed after the second treatment with identical conditions to the previous three times. General fitness parameters will be measured the same day of all the MITs to have accurate results.

#### Randomization

All subjects who consent to participation and who meet the inclusion criteria will be randomly assigned by an investigator who will not have any other interference in the clinical study; he will create a database with all the treatments through the duration of the study. Therefore, randomization will be carried out without any influence of the principal investigators. Participants will be randomly assigned to *S maxima* or placebo treatment with a 1:1 allocation according to a computergenerated random schedule stratified by site and the baseline score of the Action Arm Research Test using permuted blocks of random sizes with an online, central randomization service (TENALEA). Block sizes will not be disclosed, to ensure concealment.

#### Adherence assessments

Multiple methods will be used to assess treatment adherence including pill counting; reasons for non-compliance, and use of the capsules. Participants will return each week to receive new capsules. All treatment data will be recorded on the appropriate case report form.

### Dietary analysis

All participants will be subjected to a nutritional survey to define the daily calories required to establish a custom diet. Dietary intake will be monitored through retrospective methods including the 24 h recall (which investigates intake over a specific day), and the food frequency questionnaire (a summary of usual intake of different categories of foods). These accurate and validated techniques allow quantifying the types and quantities of foods and beverages consumed during the period of interest in the past. Dietary intake evaluations will be performed at each MIT of the study in order to record the possible variability in food consumption patterns.

# Physical exercise protocol

General health assessment and physical activity questionnaires (PAR-Q and YOU) will be conducted; this will be done to ensure that there are no physical impediments to exercise. GEx participants are going to exercise five days a week with the following protocol: between 5 and 10 min of warm-up exercise, between 20-30 min muscular endurance exercise and 20-30 minutes of aerobic exercise (cardiovascular exercise): walking, jogging, running and/or cycling. Three days a week aerobic intensities will be between 60% and 80% and two days between 70% and 90% of the maximum HR reserve, and five final minutes of stretching.

#### Sample collection and biochemical analysis

Blood samples (8 mL) will be collected before and after each MIT from the antecubital vein into ethylenediaminetetraacetic acid (EDTA) tubes after 10-12 h of

fasting, plasma from blood samples will be obtained by refrigerated centrifugation (4°C) at 5 000 g for 10 minutes. Plasma glucose TC, HDL-c, LDL-c, and TAG concentrations will be analyzed by using standard enzymatic procedures (Jas Diagnostics, Inc. Mexico) with a spectrophotometer (Genesys 10 UV; Thermo Electron Corporation, USA). Plasma will be used to measure MDA and GSH content and activity of GPx and GR according to Jimenez-Osorio *et al.* <sup>30</sup>, total antioxidant status (TAS) by 2,2-diphenyl-1-picrylhydrazyl (DPPH) technique as previously described by Koren *et al.* <sup>31</sup>, oxygen radical absorbance capacity (ORAC) following Prior *et al.* <sup>32</sup> methodology. The erythrocytes will be washed with cold 0.9% saline solution twice and are going to be used for SOD and catalase activity assays as previously described by Jimenez-Osorio *et al.* <sup>30</sup>, and plasma PON1 content will be measured by following Perez-Herrera *et al.* <sup>33</sup> methods.

#### Statistical analysis

To evaluate data distribution, normality and homoscedasticity tests on each of response variables analyzed will be conducted. In order to analyze differences between variables before and after the study and between the groups, an ANOVA test will be performed. To analyze possible associations between variables, a bivariate correlation analysis will be used. To analyze independence between variables, a multiple regression analysis will be performed. The software to use is GraphPad Prism 6.

#### **Discussion**

Cardiovascular diseases are the leading cause of mortality worldwide, with OxS. overweight, obesity, and dyslipidemias being the main risk factors. Many drugs aimed at reducing these risk factors have often collateral side effects when used, and many people often use complementary medicine instead. For this and other reasons, the pharmacological industries have focused on developing new treatment options<sup>34</sup>: S. maxima research has proven benefits to reduce CVD risk factors, isolated or in combination with systematic practice of physical exercise, mainly in animal models 9, 35, 36. This study is summarized and described in experimental design, procedures, compliance with ethical principles, and statistical analyses. Since the double-blind design, compressively described the methodology and a higher number of participants than other studies, it is expected to get a better support for the hypothesis that *S. maxima* will have hypolipidemic and antioxidant effect against intense exercise and obesity. It is noteworthy that, not every overweight or obese patient has issues with lipid metabolism, nowadays the association between the augmentation of body fat and lipid disturbances is well known <sup>37</sup>; for that reason, the primary focus of this protocol is prevention and it justifies why we do not consider dyslipidemia as an inclusion criterion; even though, they could present this condition.

247

248

249

250

251

252

253

254

255

256

257

258

259

260

261

262

263

264

265

266

267

268

269

Finally, it is known that systematic practice of exercise and a balanced diet not only favors reduction of weight in obese people, but it generally decreases cardiometabolic risks <sup>2</sup>, and thus it probably generates an increase in antioxidant capacity <sup>38</sup>; however, no studies on the metabolic oxidation decreased by

administration of *Spirulina* in people with obesity were identified. In conclusion, well-designed trials are needed to clarify the value of *S. maxima* supplementation in clinical practice <sup>39</sup>and its complementary effect with or without exercise against dyslipidemias and OxS in overweight and obesity, a fact practically unknown at this time<sup>40</sup>. The later establishes the importance of this study.

## **Competing interests**

The authors declare that they have no competing interests.

# Funding

270

271

272

273

274

275

276

277

283

- 278 This research will be funded by Programa para el Desarrollo Profesional Docente,
- SEP, México; and by Universidad Autonoma de Ciudad Juarez, Chihuahua.
- Mexico. Study design; collection, management, analysis, interpretation of data; and
- the decision to submit the results for publication will be/are all independent of the
- funders. Ultimate authority for these activities will lie with principal investigators.

# **Author affiliations**

- <sup>1</sup>Departamento de Ciencias Químico Biológicas, Instituto de Ciencias Biomédicas.
- Universidad Autónoma de Ciudad Juárez, Ciudad Juárez, Chihuahua, México.
- <sup>2</sup>Departamento de Ciencias de la Salud, Instituto de Ciencias Biomédicas.
- Universidad Autónoma de Ciudad Juárez, Ciudad Juárez, Chihuahua, México.
- <sup>3</sup>Departamento de Bioquímica, Facultad de Medicina, Universidad Nacional
- 289 Autónoma de México, Ciudad de México. <sup>4</sup>Facultad de Ciencias de la Cultura
- 290 Física, Universidad Autónoma de Chihuahua, Chihuahua, México. <sup>5</sup> Departamento

- de Biología, Facultad de Química, Universidad Nacional Autónoma de México,
- 292 Ciudad de México.

#### **Contributors**

293

300

305

All authors contributed to the development of the study protocol and to the critical revision of the paper and approved the final version. RPHT, ARJ, and JALD will be involved in patients' recruitment. MAHL and AWM will analyze the data, MAHL and MAJO will do the lipid profile analyses, RUR, ARJ and MAHL will do the body composition measurements of all patients, LARC and JPC will do all the redox status analysis.

### **Acknowledgements**

- We want to thank the Universidad Autonoma de Ciudad Juarez Institutional
  Bioethics Committee for the interest in this study, approving it and all its
  procedures. Also, we thank the Consejo Nacional de Ciencia y Tecnologia
  (CONACyT) by providing a scholarship to the first author.
  - References
- 1. WHO, World Health Organization. Fact sheet N°317. 2015. http://
   www.who.int/mediacentre/factsheets/fs317/en/. Accessed November 9<sup>th</sup> 2015.
- 2. Genest J, Frohlich J, Fodor G, McPherson R. Recommendations for the management of dyslipidemia and the prevention of cardiovascular disease: summary of the 2003 update. *CMAJ.* 2003; *169*: 921-924.

- 3. Ebbeling CB, Pawlak DB, Ludwig DS. Childhood obesity: public-health crisis,
- common sense cure. *The lancet*, 2002; 360 (9331): 473-482.
- 4. Furukawa S, Fujita T, Shimabukuro M, Iwaki M, Yamada Y, Nakajima Y,
- Shimomura I. Increased oxidative stress in obesity and its impact on
- metabolic syndrome. *Journal of Clinical Investigation*. 2004; 114 (12): 1752-
- 316 1761.
- 5. Li S, Chen W, Srinivasan SR, Bond MG, Tang R, Urbina EM, Berenson GS.
- Childhood cardiovascular risk factors and carotid vascular changes in
- adulthood: the Bogalusa Heart Study. *Jama*. 2003; 290 (17): 2271-2276.
- 6. Halliwell B, Cross CE. Oxygen-derived species: their relation to human disease
- and environmental stress. *Environmental health perspectives*. 1994; 102
- 322 Suppl 10: 5.
- 7. Schieber M, Chandel NS. ROS function in redox signaling and oxidative stress.
- 324 *Current Biology*. 2014; 24 (10): R453-R62.
- 8. Madamanchi NR, Vendrov, A, Runge MS. Oxidative stress and vascular
- disease. Arterioscler Thromb Vasc Biol. 2005; 25: 29-38.
- 9. Blé-Castillo JL, Rodriguez-Hernández A, Miranda-Zamora R, Juárez-Oropeza
- MA, Diaz-Zagoya JC. Arthrospira maxima prevents the acute fatty liver
- induced by the administration of simvastatin, ethanol and a
- hypercholesterolemic diet to mice. *Life Sci.* 2002; 70: 2665-73.
- 10. Estruch R, Ros E, Salas-Salvadó J, Covas MI, Corella D, Arós F, Martínez-
- González MA. Primary prevention of cardiovascular disease with a
- 333 Mediterranean diet. New England Journal of Medicine. 2013; 368 (14):
- 334 1279-1290.

- 11. Hoseini SM, Khosravi-Darani K, Mozafari MR. Nutritional and medical
- applications of spirulina microalgae. *Mini Rev Med Chem*; 2013. 13: 1231-7.
- 12. Chamorro G, Salazar M, Favila L, Bourges H. Pharmacology and toxicology of
- 338 Spirulina alga. *Rev Invest Clin.* 1995; 48: 389-99.
- 13. Iwata K, Inayama T, Kato T. Effects of Spirulina platensis on plasma lipoprotein
- lipase activity in fructose-induced hyperlipidemic rats. *J Nutr Sci Vitaminol*
- 341 (*Tokyo*). 1990; 36: 165-71.
- 14. Riss J, Décordé K, Sutra T, Delage M, Baccou J, Jouy N. Phycobiliprotein C-
- phycocyanin from Spirulina platensis is powerfully responsible for reducing
- oxidative stress and NADPH oxidase expression induced by an atherogenic
- diet in hamsters. *J Agric Food Chem.* 2007; 55: 7962-7967.
- 15. Torres-Duran PV, Ferreira-Hermosillo A, Juarez-Oropeza MA. Antihyperlipemic
- and antihypertensive effects of Spirulina maxima in an open sample of
- Mexican population: a preliminary report. *Lipids Health Dis.* 2007; 6: 33.
- 16. Pérez IP, Álvarez FV, López PM, Jiménez FP, Galán AM, Lenguas JAC, López
- EG. Control de la colesterolemia en España, 2000. Un instrumento para la
- prevención cardiovascular. Revista Española de Cardiología. 2000; 53 (6):
- 352 815-837.
- 17. Fisher-Wellman K, Bloomer RJ. Acute exercise and oxidative stress: a 30 year
- history. *Dynamic Medicine*. 2009; 8 (1): 1.
- 18. Morillas-Ruiz JM, García JV, López FJ, Vidal-Guevara ML, Zafrilla P. Effects of
- polyphenolic antioxidants on exercise-induced oxidative stress. *Clinical*
- 357 *Nutrition*. 2006; 25 (3): 444-453.

- 19. Aoi W, Naito Y, Yoshikawa T. Role of oxidative stress in impaired insulin signaling associated with exercise-induced muscle damage. *Free Radical Biology and Medicine*. 2013; 65: 1265-1272.
- 20. Gomez-Cabrera MC, Domenech E, Viña J. Moderate exercise is an
   antioxidant: upregulation of antioxidant genes by training. *Free Radical Biology and Medicine*. 2008; 44 (2): 126-131.
- 21. Savini I, Catani MV, Evangelista D, Gasperi V, Avigliano L. Obesity-associated oxidative stress: strategies finalized to improve redox state. *International journal of molecular sciences*. 2013; 14, (5): 10497-10538.
- 22. Gammone MA, Gemello E, Riccioni G, D'Orazio, N. Marine bioactives and potential application in sports. *Marine drugs*. 2014; 12(5), 2357-2382.
- 23. Gammone MA, D'Orazio N. Anti-obesity activity of the marine carotenoid fucoxanthin. *Marine drugs*. 2015; 13(4), 2196-2214.
- 24. Upasani CD, Khera A, Balaraman R. Effect of lead with vitamin E, C, or
   Spirulina on malondialdehyde, conjugated dienes and hydroperoxides in
   rats. *Indian J Exp Biol.* 2001; 39: 70–74.
- 25. Nagaoka S, Shimizu K, Kaneko H, Shibayama F, Morikawa K, Kanamaru Y,
   Kato T. A novel protein C-phycocyanin plays a crucial role in the
   hypocholesterolemic action of Spirulina platensis concentrate in rats. *J Nutr*.
   2005; 135: 2425-30.
- 26. Thaakur SR, Jyothi B. Effect of Spirulina maxima on the haloperidol induced tardive dyskinesia and oxidative stress in rats. *J Neural Transm*. 2007; 114: 1217–1225.

- 27. Stewart A, Marfell-Jones M, Olds T, de Ridder H. International standards for
- anthropometric assessment. 2011: ISAK: Lower Hutt, New Zealand
- 28. Mao TK, Water JVD, Gershwin ME. Effects of a Spirulina-based dietary
- supplement on cytokine production from allergic rhinitis patients. *Journal of*
- 385 *Medicinal Food*. 2005; 8(1), 27-30.
- 29. Faul F, Erdfelder E, Lang AG, Buchner A. G\* Power 3: A flexible statistical
- power analysis program for the social, behavioral, and biomedical sciences.
- 388 Behavior research methods. 2007; 39(2), 175-191.
- 30. Jiménez-Osorio, AS, Picazo, A, González-Reyes, S, Barrera-Oviedo, D,
- Rodríguez-Arellano, ME, Pedraza-Chaverri, J. Nrf2 and redox status in
- prediabetic and diabetic patients. *International journal of molecular sciences*.
- 392 2014; 15(11), 20290-20305.
- 393 31. Koren E, Kohen R, Ginsburg I. Polyphenols enhance total oxidant-scavenging
- capacities of human blood by binding to red blood cells. *Experimental*
- 395 Biology and Medicine. 2010; 235(6), 689-699.
- 396 32. Prior, RL, Hoang, HA, Gu, L, Wu, X, Bacchiocca, M, Howard, L, Jacob, R.
- Assays for hydrophilic and lipophilic antioxidant capacity (oxygen radical
- absorbance capacity (ORACFL)) of plasma and other biological and food
- samples. Journal of Agricultural and Food Chemistry. 2003; 51(11), 3273-
- 400 3279.
- 401 33. Pérez-Herrera, N. May-Pech, C. Hernández-Ochoa, I. Castro-Mañé, J. Rojas-
- 402 García, E, Borja-Aburto, VH, Quintanilla-Vega, B. PON1Q192R

- polymorphism is associated with lipid profile in Mexican men with Mayan ascendancy. *Experimental and molecular pathology*. 2008; 85(2), 129-134.
- 34. Banach M, Stulc T, Dent R, Toth PP. Statin non-adherence and residual
   cardiovascular risk: There is need for substantial improvement. *International Journal of Cardiology*. 2016; 225, 184-196.
- 35. Cheong SH, Kim MY, Sok DE, Hwang SY, Kim JH, Kim HR, Kim MR. Spirulina prevents atherosclerosis by reducing hypercholesterolemia in rabbits fed a high-cholesterol diet. *J Nutr Sci Vitaminol (Tokyo)*. 2010; 56: 34-40.
- 36. Moura LP, Puga GM, Beck WR, Teixeira IP, Ghezzi AC, Silva GA, Mello MA.
   Exercise and spirulina control non-alcoholic hepatic steatosis and lipid
- profile in diabetic Wistar rats. *Lipids Health Dis.* 2011; 10: 77.
- 37. Ugwuja EI, Ogbonna NC, Nwibo AN, Onimawo IA. Overweight and obesity,
  lipid profile and atherogenic indices among civil servants in Abakaliki, south
  eastern Nigeria. *Annals of medical and health sciences research*. 2013;
  3(1), 13-18.
- 38. Fenster CP, Weinsier RL, Darley-Usmar VM, Patel RP. Obesity, aerobic
  exercise, and vascular disease: the role of oxidant stress. *Obesity research*.
  2002; *10*(9): 964-968.
- 39. Serban MC, Sahebkar A, Dragan S, Stoichescu-Hogea G, Ursoniu S, Andrica
  F, Banach M. A systematic review and meta-analysis of the impact of
  Spirulina supplementation on plasma lipid concentrations. *Clinical nutrition*.
  2016; 35(4), 842-851.

- 40. Hernández-Lepe MA, Wall-Medrano A, Juárez-Oropeza MA, Ramos-Jiménez,
- A, Hernández-Torres RP. Spirulina y su efecto hipolipemiante y antioxidante
- en humanos: una revisión sistemática. *Nutr Hosp.* 2015; 32(2), 494-500.



**Figure 1.** Experimental design for independent and synergistic effect of *Spirulina* maxima and exercise. Same color means the same group of participants.



**Figure 2.** Design of maximum intensity tests. ↓ indicates the interval at which the resistance will be increased; in addition, physical perceived effort, heart rate, and capillary blood samples will be measured.